## Impact of Self-Awareness in Stress, Burnout, Self-Compassion and Compassion in medical students

## 096/2019

## 1 June 2020 version



## RESEARCH PROTOCOL

Title:

Impact of Self-Awareness in Stress, Burnout, Self-Compassion and Compassion in medical students

INTRODUCTION: It has been proven that the training of future physicians generates high levels of stress, from the need to assimilate a lot of knowledge in a short time to the anxiety of anticipating the practical profession. This reality has been translated into increasing burnout rates in medical students, whose physical, psychological and behavioral impact translates into repercussions on the quality of life of students and on their role as physicians and on the patients themselves. It therefore becomes an ethical duty to find and develop tools for stress management and burnout prevention. Currently, there are several studies that address individual, organizational, and combined strategies. However, few have sought to relate self-knowledge as a protective factor against burnout inducers. According to Rispail (2003) and Cunha et al. (2013), self-knowledge involves what we think of ourselves implying a self-evaluation of limits, fears, insecurities, and vulnerability, but also of potentialities. In Portugal, it was tried to understand its protective role against burnout in intensive care units, but not in medical students. In 2019, we conducted a pilot study of this trial, which we now intend to extend to a larger sample.

OBJECTIVES: To understand if the promotion of self-awareness in medical students based on the Enneagram of Personalities tool has an impact on levels of stress, burnout, and quality of life in this population, as well as on self-compassion and compassion, promoting awareness of its importance and possible application in medical schools.

METHODS: First, an online outreach will be conducted to solicit volunteers within the medical students. After acquiring a randomly selected representative sample within the volunteers, a randomized controlled clinical trial will be conducted, where the intervention will consist of a course, guided by specialized trainers, in which self-knowledge skills will be developed and self-knowledge skills and training in communication and empathy. This course will be divided into 3 sessions: in a first, a theoretical introduction is given, where the Personality Enneagram is addressed; in the second, the p

articipants will try to apply what they have learned to self-knowledge and seek ways of growth and stress management; finally, they will be confronted with practical situations similar to those they will face in the future as doctors, applying the previous knowledge. The groups will have to answer 2 online questionnaires with 6 scales, before and after the intervention and 9 months later. The results obtained will be subject to descriptive and inferential descriptive and inferential statistical analysis.

- 1. Ishak W, Nikravesh R, Lederer S, Perry R, Ogunyemi D, Bernstein C. Burnout in medical students: a systematic review. Clin Teach. 2013;10(4):242-5.
- 2. Novack DH, Epstein RM, Paulsen RH. Toward creating physician-healers: fostering medical students' selfawareness, personal growth, and well-being. Acad Med. 1999;74(5):516-20.
- 3. Shiralkar MT, Harris TB, Eddins-Folensbee FF, Coverdale JH. A systematic review of stress-management programs for medical students. Acad Psychiatry. 2013;37(3):158-64.

Authors:

ANA CAROLINA MONTEIRO MARTINHO INÊS ROSENDO CARVALHO E SILVA LILIANA RUTE ANTONIO CONSTANTINO